CLINICAL TRIAL: NCT00573599
Title: Prochlorperazine vs Imitrex for Acute Migraine in the Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit participants
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06-050
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Migraine Headache
Keywords: Migraine; Emergency; imitrex; prochlorperazine; Acute Migraine Headache in the Emergency Department
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — Prochlorperazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): prochlorperazine and benadryl IV, saline subQ
  Interventions: Drug: prochlorperazine and benadryl IV
- 2 (Active Comparator): imitrex SubQ, saline IV
  Interventions: Drug: Imitrex SubQ, saline IV

INTERVENTIONS:
Drug: prochlorperazine and benadryl IV — prochlorperazine and benadryl IV, saline subQ
  Arms: 1
Drug: Imitrex SubQ, saline IV — Imitrex SubQ, saline IV
  Arms: 2

SUMMARY:
ED patients with acute migraine will be randomized to either prochlorperazine and Bendaryl OR imitrex. VAS for pain will be monitored, along with side effects. Primary outcome measure is improvement in pain scales between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Acute migraine headache

Exclusion Criteria:

* Pregnant
* Hypertension
* Chest pain
* < 18
* Allergy to any of the meds

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Difference in pain measured by VAS | 80 min

SECONDARY OUTCOMES:
Degree of sedation, nausea, akathisia | 80 min

CONTACTS AND LOCATIONS:
Overall Officials: Frank Gutierrez, MD, Principal Investigator — US Navy
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States